CLINICAL TRIAL: NCT02750657
Title: Comprehensive Molecular Characterization of Advanced Pancreatic Ductal Adenocarcinomas (PDAC) for Better Treatment Selection: A Prospective Study
Brief Title: Study of Changes and Characteristics of Genes in Patients With Pancreatic Cancer for Better Treatment Selection
Acronym: COMPASS
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: COMPASS-001
Record Dates: First submitted 2016-01-19; First posted 2016-04-25 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Pancreatic Ductal
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: * Fresh tumor tissue biopsy samples
  * Archival tumor tissue samples
  * Whole blood samples
  * Plasma samples
  * Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with advanced pancreatic ductal adenocarcinoma
  Interventions: Genetic: Molecular Profiling

INTERVENTIONS:
Genetic: Molecular Profiling — Whole Genome Sequencing

SUMMARY:
Researchers are looking for better ways of understanding and treating pancreatic cancer. The purpose of this study is to see how useful it is to look for changes and characteristics in your genes (molecules that contain instructions for the development and functioning of the cells) and the genes within the tumour. These characteristics may be useful in choosing treatments for patients in the future. Changes (mutations) in genes have been shown to be an important characteristic in cancers. Looking at differences in genes in patients with advanced pancreatic ductal adenocarcinomas and comparing this information with response to their initial chemotherapy treatment may help to learn which treatments may be better for certain patients after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological or radiological diagnosis of locally advanced or metastatic pancreatic ductal adenocarcinoma. Patients with borderline resectable disease are not eligible.
* Patient must have a tumor lesion that is amenable to a core needle biopsy.
* Patients must have a measurable lesion by RECIST 1.1 in addition to the lesion that is going to be biopsied.
* Patients must be fit enough to safely undergo a tumor biopsy.
* Age 18 years or older.
* Eastern Cooperative Group (ECOG) performance status of 1 or less.
* Life expectancy of greater than 90 days.
* Patients must have normal organ and marrow function
* Patients must undergo systemic treatment with m-FOLFIRINOX or nab-paclitaxel as a first line standard systemic palliative treatment or combination treatment with m-FOLFIRINOX or nab-paclitaxel with or without other investigational agents within a clinical trial as a first line palliative treatment.
* Ability to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patients with one or more contraindications to tumor biopsy.
* Patients who have prior systemic treatment (chemotherapy or any other anti-cancer agent) in advanced setting.
* Patients who are currently on anti-cancer treatment including chemotherapy.
* Patients with known brain metastases.
* Patients with advanced PDAC who are going to be treated with gemcitabine monotherapy in advanced setting.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced or metastatic pancreatic ductal adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2025-08 (Actual); Study Completion 2025-08 (Actual)

PRIMARY OUTCOMES:
The feasibility of prospectively identifying subgroups of patients with advanced PDAC who have distinct genomic characteristics for better treatment selection while undergoing 1st-line chemotherapy using next generation sequencing. | 8 weeks

SECONDARY OUTCOMES:
Disease control rate achieved by m-FOLFIRINOX | 5 years
Disease control rate achieved by nab-paclitaxel | 5 years
Duration of response defined as the interval between the first date of complete response or partial response and the earliest date of disease progression or death due to any cause to m-FOLFIRINOX | 5 years
Duration of response defined as the interval between the first date of complete response or partial response and the earliest date of disease progression or death due to any cause to nab-paclitaxel. | 5 years
Progression free survival defined as the interval between the date of registration and the earliest date of disease progression or death due to any cause of patients treated with m-FOLFIRINOX. | 5 years
Progression free survival defined as the interval between the date of registration and the earliest date of disease progression or death due to any cause of patients treated with nab-paclitaxel. | 5 years
Overall survival defined as the interval between the date of registration and the date of death of patients treated with m-FOLFIRINOX | 5 years
Overall survival defined as the interval between the date of registration and the date of death of patients treated with nab-paclitaxel. | 5 years
Correlation between tumor genomic characteristics and m-FOLFIRINOX response using next generation sequencing. | 5 years
Correlation between tumor genomic characteristics and nab-paclitaxel response using the next generation sequencing. | 5 years
Percentage of patients with germline BRCA, PALB2 and ATM mutations who might benefit from a personalized treatment strategy such as combination of cisplatin and a PARP inhibition. | 5 years
Percentage of patients with somatic DSBR deficiency who might benefit from a personalized treatment strategy such as combination of cisplatin and a PARP inhibitor. | 5 years
Percentage of patients who might benefit from immunotherapy (patients with smoking genomic signatures, patients with a hypermutated phenotype, patients with mismatch repair deficiency and patients with tumor neo-antigen expression). | 5 years
Percentage of patients with rare but targetable somatic mutations. | 5 years
Difference in disease control rate between patients with tumor smoking signature and those without. | 5 years
Difference in overall survival between patients with tumor smoking signature and those without. | 5 years
Correlation with tumor molecular characteristics and toxicities to treatment using next generation sequencing. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J. Knox, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (4):
- Canada (4):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Derived] Karasinska JM, Topham JT, Kalloger SE, Jang GH, Denroche RE, Culibrk L, Williamson LM, Wong HL, Lee MKC, O'Kane GM, Moore RA, Mungall AJ, Moore MJ, Warren C, Metcalfe A, Notta F, Knox JJ, Gallinger S, Laskin J, Marra MA, Jones SJM, Renouf DJ, Schaeffer DF. Altered Gene Expression along the Glycolysis-Cholesterol Synthesis Axis Is Associated with Outcome in Pancreatic Cancer. Clin Cancer Res. 2020 Jan 1;26(1):135-146. doi: 10.1158/1078-0432.CCR-19-1543. Epub 2019 Sep 3. PMID 31481506
- [Derived] Aung KL, Fischer SE, Denroche RE, Jang GH, Dodd A, Creighton S, Southwood B, Liang SB, Chadwick D, Zhang A, O'Kane GM, Albaba H, Moura S, Grant RC, Miller JK, Mbabaali F, Pasternack D, Lungu IM, Bartlett JMS, Ghai S, Lemire M, Holter S, Connor AA, Moffitt RA, Yeh JJ, Timms L, Krzyzanowski PM, Dhani N, Hedley D, Notta F, Wilson JM, Moore MJ, Gallinger S, Knox JJ. Genomics-Driven Precision Medicine for Advanced Pancreatic Cancer: Early Results from the COMPASS Trial. Clin Cancer Res. 2018 Mar 15;24(6):1344-1354. doi: 10.1158/1078-0432.CCR-17-2994. Epub 2017 Dec 29. PMID 29288237